CLINICAL TRIAL: NCT03934008
Title: An Observational Study to Analyze the Effectiveness of a Motivational Interviewing-based Decision Tool to Address Vaccination Hesitancy in Children
Brief Title: Motivational Interviewing and Vaccine Hesitancy in Children
Acronym: MOTIVE
Status: Completed | Type: Observational
Sponsor: Cedarville University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Rocking Horse Community Health Center (Unknown)
Responsible Party: Principal Investigator, Justin Cole, Assistant Professor and Interim Chair of Pharmacy Practice, Cedarville University
Other Study IDs: IRB #997
Record Dates: First submitted 2019-03-22; First posted 2019-05-01 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Vaccine Hesitancy
Keywords: Motivational Interviewing; Pediatrics
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Historical Control Group: All pediatric patients 0-6 years of age seen in the clinic within one year prior to the start of the intervention period
- Post-Intervention Group: All pediatric patients 0-6 years of age seen in the clinic for one year following the implementation of the motivational interviewed based tool
  Interventions: Other: MOtivational interviewing Tool to Improve Vaccine AdherencE (MOTIVE)

INTERVENTIONS:
Other: MOtivational interviewing Tool to Improve Vaccine AdherencE (MOTIVE) — The MOTIVE tool incorporates the principles of motivational interviewing (MI) and provides a flowchart approach in which parental health beliefs have a corresponding MI-based strategy to further explore and/or address the hesitancy. The tool was developed from interviews with pediatricians and pediatric pharmacists, a review of the literature focusing on vaccine health beliefs, and the Parent Attitudes about Childhood Vaccines (PACV) Survey Tool. The tool was reviewed by multiple providers and feedback was provided on its usability in clinical practice when interacting with vaccine-hesitant parents and/or caregivers. The tool was then modified based on this feedback. Pediatric providers will complete four educational sessions on vaccine hesitancy, MI, and the use of the MOTIVE tool in clinical practice prior implementation.
  Groups: Post-Intervention Group

SUMMARY:
This study will assess the effectiveness of a motivational interviewing-based tool in addressing vaccine hesitancy expressed by parents or caregivers of children.

DETAILED DESCRIPTION:
In order for vaccines to be effective and protect communities from diseases, a large majority of individuals need to be vaccinated to protect those who do not respond to the vaccine and those who cannot be vaccinated. While vaccine hesitancy has been noted as a growing problem among parents, there are few evidence-based strategies for providers to utilize to discuss vaccination with these parents. Therefore, there is a critical need to develop effective communication tools to increase parental confidence in vaccines. A tool based on the principles of motivational interviewing (a goal-oriented, collaborative counseling style) may be effective in addressing this need. Thus, the aim of this study is to determine the impact of a motivational interviewing-based (MI-based) tool on pediatric vaccination rates through assessment of changes in the percentage of patients achieving the goal of completion of all recommended doses in children 6 years of age and younger. Secondary aims include determining the impact of the motivational-interviewing based tool on parental health beliefs regarding vaccines and the impact of the training on provider knowledge and confidence in using motivational interviewing.

ELIGIBILITY:
Inclusion Criteria (primary outcome):

* Patients 0-6 years of age
* Seen in the Rocking Horse Community Center by a pediatric provider during the baseline or study period

Inclusion Criteria (secondary parental health belief outcomes):

* Parents/caregivers (1) ≥18 years old
* Read English
* Have at least one child ≤6 years of age

Inclusion Criteria (secondary provider outcomes): All providers who interact with pediatric patients in the Rocking Horse Community Center who

* Complete the training
* Implement the MOTIVE tool in practice

Ages: 0 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients, parents/caregivers, and providers at the Rocking Horse Community Center
Sampling Method: Non-Probability Sample
Enrollment: 4191 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
The percentage of children 0-6 years of age receiving all recommended doses of the core vaccine series | Change from baseline at 12 months post intervention implementation
  The percentage of eligible patients presenting for care at Rocking Horse Community Center who receive all doses of the core immunization series (HepB, DTaP, Hib, PCV13, IPV, MMR, VAR, Hep A) for the patient's age according to the Advisory Committee on Immunization Practices (ACIP) and Centers for Disease Control (CDC) Immunization Schedule during the intervention year compared to the same percentage in the control group over the previous year.
The percentage of children 0-6 years of age receiving all recommended vaccines doses | Change from baseline at 12 months post intervention implementation
  The percentage of eligible patients presenting for care at Rocking Horse Community Center who receive all doses (including rotavirus and influenza) of recommended vaccines according to the ACIP/CDC Immunization Schedule during the intervention year compared to the same percentage in the control group over the previous year.
The percentage of children 0-6 years of age receiving appropriate influenza vaccination | Change from baseline at 12 months post intervention implementation
  The percentage of eligible patients presenting for care at Rocking Horse Community Center who receive appropriate influenza vaccination according to the ACIP/CDC Immunization Schedule during the intervention year compared to the percentage in the control group over the previous year.
Number of deferred vaccine doses | Change from baseline at 12 months post intervention implementation
  Number of deferred vaccine doses per 100 patients during the intervention year compared to the number of deferred vaccine doses in the control group over the previous year.

SECONDARY OUTCOMES:
Parental attitude towards vaccines (PACV total score) | Change from baseline at post-encounter assessment (within 24 hours of receiving MI-based intervention)
  The difference in Parental Attitudes about Childhood Vaccines (PACV) total score (range 0-100, with higher scores indicating greater hesitancy) in parents who have answered yes to items 3 and 4 in the pre-survey population compared to those who receive the MI-based intervention.
Provider knowledge of utilizing motivational interviewing to address vaccine hesitancy | Change from baseline at 2 months after the provider training period is completed
  The change in the Knowledge subscale (5 items, range 0-5, with higher scores indicating greater knowledge) of the Motivational Interviewing Provider Scale.
Provider confidence in utilizing motivational interviewing to address vaccine hesitancy | Change from baseline at 2 months after the provider training period is completed
  The change in the Confidence subscale (range 16-96, with higher scores indicating greater confidence) of the Motivational Interviewing Provider Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Justin W Cole, PharmD, Principal Investigator — Cedarville University School of Pharmacy
Locations (1):
- Rocking Horse Community Heath Center, Springfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cole JW, M H Chen A, McGuire K, Berman S, Gardner J, Teegala Y. Motivational interviewing and vaccine acceptance in children: The MOTIVE study. Vaccine. 2022 Mar 15;40(12):1846-1854. doi: 10.1016/j.vaccine.2022.01.058. Epub 2022 Feb 10. PMID 35153096